CLINICAL TRIAL: NCT01976442
Title: Impact of Washed Transfusions in Adult Patients With Acute Myeloid or Lymphoid Leukemia
Brief Title: Use of Saline-Washed Platelet and Red Cell Transfusions in Adult Acute Leukemia
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Neil Blumberg, Professor, University of Rochester
Other Study IDs: URMC RSRB00035034
Record Dates: First submitted 2013-10-16; First posted 2013-11-05 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Lymphoblastic, Acute
Keywords: Leukemia; Transfusion
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether a novel standard of care protocol, washing red cell and platelet transfusions for younger patients with acute leukemia, has yielded improved clinical outcomes at Strong Memorial Hospital (Rochester, New York, USA). This standard of care was implemented based upon an earlier randomized trial (BMC Blood Disorders. 2004 Dec 10;4(1):6) The comparator will be historical controls from the medical literature.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether a novel standard of care protocol, washing red cell and platelet transfusions for younger patients with acute leukemia, has yielded improved clinical outcomes at Strong Memorial Hospital (Rochester, New York, USA). This standard of care was implemented based upon an earlier randomized trial (BMC Blood Disorders. 2004 Dec 10;4(1):6) The comparator will be historical controls from the medical literature. Key outcomes will be treatment related mortality (deaths at 30, 60 and 100 days) and three year survival.

ELIGIBILITY:
Inclusion Criteria:

* previously untreated patients with a diagnosis of acute leukemia between the ages of 0 and 50 (AML) and 18 and 50 (ALL)

Exclusion Criteria:

* all other patients

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population is comprised of 98 men and women who were both diagnosed and treated for Acute Myeloid Leukemia or Acute Lymphoid Leukemia at Strong Memorial Hospital, a tertiary medical center located in Rochester, NY, USA. All of these patients received washed red cell and platelet transfusions as part of the hospital's standard protocol for patients with acute leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Blumberg, M.D., Principal Investigator — University of Rochester Medical Center, School of Medicine and Dentistry
Locations (1):
- Strong Memorial Hospital (University of Rochester Medical Center), Rochester, New York, United States

REFERENCES:
- [Background] Blumberg N, Heal JM, Rowe JM. A randomized trial of washed red blood cell and platelet transfusions in adult acute leukemia [ISRCTN76536440]. BMC Blood Disord. 2004 Dec 10;4(1):6. doi: 10.1186/1471-2326-4-6. PMID 15588315

RESULTS

PARTICIPANT FLOW:
Groups:
- Washed: Washed red blood cell transfusions given to all patients with acute myeloid leukemia.
- Unwashed: Transfusions of red cells were not washed before transfusion into the acute myeloid leukemia patient.
Period: Overall Study
Arm/Group | Washed | Unwashed
Started | 69 | 31
Completed | 69 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Washed | Unwashed | Total
Number analyzed (Participants) | 69 | 31 | 100
Age, Continuous [Mean (Full Range); unit: years] | 40 [1 to 50] | 30 [2 to 49] | 35 [1 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 18 | 64
  Male | 23 | 13 | 36
Region of Enrollment [Number; unit: participants]
  United States | 69 | 31 | 100

OUTCOME MEASURES:

1. Primary Outcome: Survial Rate at 30 Days
Description: The percentage of patients who were alive at 30 days after transfusion.
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | Washed | Unwashed
Number analyzed (Participants) | 69 | 31
percentage of participants | 100 | 97

2. Primary Outcome: Survial Rate at 60 Days
Description: The percentage of patients who were alive at 60 days after transfusion.
Time Frame: 60 days
Measure: Number; unit: percentage of participants
Arm/Group | Washed | Unwashed
Number analyzed (Participants) | 69 | 31
percentage of participants | 97 | 94

3. Primary Outcome: Survial Rate at 100 Days
Description: The percentage of patients who were alive at 100 days after transfusion.
Time Frame: 100 days
Measure: Number; unit: percentage of participants
Arm/Group | Washed | Unwashed
Number analyzed (Participants) | 69 | 31
percentage of participants | 96 | 87

4. Primary Outcome: Survial Rate at 5 Years
Description: The percentage of patients who were alive at 5 years after transfusion.
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Washed | Unwashed
Number analyzed (Participants) | 69 | 31
percentage of participants | 55 | 39

ADVERSE EVENTS:
Description: Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Washed | Unwashed
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This is a cohort study and thus has limits as to confounding and bias. However, it reproduces the results of a previous single center randomized trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No